CLINICAL TRIAL: NCT00692081
Title: A Randomized Controlled Trial of a Social Competence Group Training for Adolescents With Borderline Intellectual Functioning
Brief Title: Social Competence Training for Adolescents With Borderline Intellectual Functioning
Acronym: SCT-ABI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UNIVULM
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Mental Disorders
Keywords: adolescents; borderline intellectual functioning; social competence training; vocational training; group intervention; cognitive behavioral therapy; Adolescents with borderline intellectual functioning
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): 8 group sessions social competence training (CBT)
  Interventions: Behavioral: Social competence training
- B (Active Comparator): special vocational training as usual
  Interventions: Behavioral: Special vocational training

INTERVENTIONS:
Behavioral: Social competence training — 8 group sessions multi-modal social competence training, 2-4 hours each, 2 trainers, 6-10 participants
  Arms: A
Behavioral: Special vocational training — as provided in German special centres for vocational training
  Arms: B

SUMMARY:
Emotional and behavioural problems as well as a lack of social competence are supposed to be common phenomena in adolescents with borderline intellectual functioning, consequently impairing their social and vocational integration. Considering the lack of evaluated group interventions for this population, a cognitive-behavioural training is developed and its effectiveness is examined in a population of students attending special vocational schools.

77 adolescents with borderline intelligence are enrolled participated in the study. They are randomized either to the intervention group, who received 9 group sessions over a period of 3 months additionally to the standard vocational training (Social Competence Training for Adolescents with Borderline Intelligence, SCT-ABI) or to the control group who received only the standard vocational training. Outcome measures at the end of the intervention and at a 6-months follow-up assessment comprise self-reports, caregiver-reports, and behavioural observations of cognitive, emotional, and behavioural factors of social competence.

ELIGIBILITY:
Inclusion Criteria:

* age 16 - 23 years
* participating in special vocational training program
* elevated scores in a screening measure of behavioral/emotional disorders (CBCL or YSR T>59)

Exclusion Criteria:

* major psychiatric disorder (psychosis, major depression, substance abuse)

Ages: 16 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 77 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lutz Goldbeck, Ph.D., Principal Investigator — University Ulm

REFERENCES:
- [Derived] Nestler J, Goldbeck L. A pilot study of social competence group training for adolescents with borderline intellectual functioning and emotional and behavioural problems (SCT-ABI). J Intellect Disabil Res. 2011 Feb;55(2):231-41. doi: 10.1111/j.1365-2788.2010.01369.x. Epub 2011 Jan 4. PMID 21199047